CLINICAL TRIAL: NCT02256748
Title: A Study to Evaluate the Effect of Multiple Doses of 500 mg of BIRT 2584 XX Tablets on the Pharmacokinetic Parameters of Midazolam in Healthy Male Volunteers
Brief Title: Study to Evaluate the Effect of Multiple Doses of BIRT 2584 XX Tablets on the Pharmacokinetic Parameters of Midazolam in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1206.9
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

ARMS (1):
- BIRT 2584 XX + Midazolam (Experimental): BIRT 2584 XX: Multiple doses for 12 days (bid on days 1 and 2, qd from days 3 to 12)
  Midazolam: Administration on days -2, 1, 3, and 12
  Interventions: Drug: BIRT 2584 XX; Drug: Midazolam

INTERVENTIONS:
Drug: BIRT 2584 XX
Drug: Midazolam

SUMMARY:
The objective of the study was to investigate the effect of BIRT 2584 XX and its metabolite BI 610100 when BIRT 2584 XX is administered as a tablet to near steady state in estimated high therapeutic dose on the pharmacokinetics (PK) of midazolam, a probe substrate for CYP3A4. The PK of midazolam was measured before dosing of BIRT 2584 XX, after a single dose of BIRT 2584 XX and after repeated doses of BIRT 2584 XX for 3 and 12 days

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of the screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age ≥ 18 and ≤ 55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding during the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hematological, oncological, or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Relevant history of orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) considered relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (greater than 24 hours) (less than 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial (less than 10 days prior to study drug administration or expected during the trial)
* Participation in another trial with an investigational drug (less than 2 months prior to administration or expected during trial)
* Smoker (more than 10 cigarettes/day or more than 3 cigars/day or more than 3 pipes/day)
* Alcohol abuse (more than 60 g of ethanol per day)
* Drug abuse
* Blood donation or loss greater than 400 mL (less than 1 month prior to administration or expected during the trial)
* Clinically relevant laboratory abnormalities

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ of midazolam (area under the concentration-time curve of midazolam in plasma over the time interval from 0 extrapolated to infinity) | up to 13 days
Cmax of midazolam (maximum concentration of midazolam in plasma) | up to 13 days
AUC0-∞ of 1'-hydroxymidazolam (area under the concentration-time curve of 1'-hydroxymidazolam in plasma over the time interval from 0 extrapolated to infinity) | up to 13 days
Cmax of 1'-hydroxymidazolam (maximum concentration of 1'-hydroxymidazolam in plasma) | up to 13 days
AUC0-∞ ratio of 1'-hydroxymidazolam to midazolam | up to 13 days

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analytes in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 13 days
tmax (time from dosing to the maximum concentration of the analytes in plasma) | up to 13 days
λz (terminal rate constant of the analytes in plasma) | up to 13 days
t1/2 (terminal half-life of the analytes in plasma) | up to 13 days
MRTpo (mean residence time of the analytes in the body after po administration) | up to 13 days
CL/F (apparent clearance of the analytes in the plasma after extravascular administration) | up to 13 days
Vz/F (apparent volume of distribution during the terminal phase following an extravascular dose) | up to 13 days
Pre-dose levels of BIRT 2584 XX and BI 610100 | days 1, 3 and 12
Number of subjects with abnormal findings in physical examination | up to 29 days
Number of subjects with abnormal changes in laboratory parameters | up to 29 days
Number of subjects with clinically significant changes in 12-lead ECG | up to 29 days
Number of subjects with clinically significant changes in vital signs | up to 29 days
  Pulse rate, systolic, and diastolic blood pressure
Number of subjects with adverse events | up to 44 days
Assessment of tolerability by investigator on a 4-point scale | Day 29